CLINICAL TRIAL: NCT00086580
Title: A Phase III Randomized Trial to Evaluate the Efficacy and Safety of Second-Line Therapy With Fludarabine Plus Alemtuzumab vs. Fludarabine Alone in Patients With B-Cell Chronic Lymphocytic Leukemia
Brief Title: Fludarabine (Fludara®) Plus Alemtuzumab (CAMPATH®, MabCampath®) vs Fludarabine Alone in B-Cell Chronic Lymphocytic Leukemia (B-CLL) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAM314; 2004-000149-39 (EudraCT Number)
Record Dates: First submitted 2004-07-06; First posted 2004-07-08 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine phosphate; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Arm (FluCAM) (Experimental)
  Interventions: Biological: FluCAM [Fludara + Campath]
- Fludarabine Alone (Active Comparator)
  Interventions: Biological: fludarabine phosphate

INTERVENTIONS:
Biological: FluCAM [Fludara + Campath] — Phase A: Escalating Doses of alemtuzumab (Campath) Alone
  Day 1: alemtuzumab 3 mg intravenously (IV) over 2 hours.
  Day 2: alemtuzumab 10 mg IV over 2 hours if 3 mg was tolerated, else repeat 3 mg daily until tolerated.
  Day 3: alemtuzumab 30 mg IV over 2 hours if 10 mg was tolerated, else repeat 10 mg daily until tolerated.
  Participants were allowed 3-14 days to escalate to 30 mg. Once 30 mg was tolerated, the participant had to begin Phase B within 7 days.
  Phase B: FluCAM
  Cycle 1: Days 1,2,3 fludarabine phosphate administered at 30 mg/m^2 over 30 minutes IV, followed within 1 hour by alemtuzumab 30 mg IV over 2 hours. A similar schedule is set for Cycles 2 through 6; duration of alemtuzumab infusions vary from 2-6 hours. Each 28-day period is 1 cycle. Fludarabine phosphate dosage is based on participants' body surface area at the beginning of each cycle. FluCAM administered up to a maximum of 6 cycles, based upon participants' response to therapy and toxicity.
  Other Names: alemtuzumab; fludarabine phosphate; Fludara; Campath
  Arms: Combination Arm (FluCAM)
Biological: fludarabine phosphate — Fludarabine phosphate (Fludara) is administered at a dose of 25 mg/m^2 IV over 15 to 30 minutes daily for 5 consecutive days (days 1 through 5) every 28 days (per package instructions). Each 28-day period is 1 cycle. The dose of fludarabine phosphate will be based on the participant's body surface area as calculated at the beginning of each cycle. Participants treated with fludarabine phosphate up to a maximum of 6 cycles, based upon their response to therapy and toxicity.
  Other Names: Fludara
  Arms: Fludarabine Alone

SUMMARY:
This is a Phase 3, prospective, multicenter, open-label, randomized, controlled study to evaluate and compare the efficacy and safety of fludarabine plus alemtuzumab versus fludarabine alone as second-line therapy for patients with relapsed or refractory B-cell chronic lymphocytic leukemia (B-CLL). Patients who meet all eligibility criteria and sign the informed consent document may be entered on the study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of B-cell chronic lymphocytic leukemia (B-CLL); according to the National Cancer Institute Working Group (NCI WG) criteria.
* Relapsed or refractory disease after 1 prior regimen except patients who were refractory to (i.e., progressed on) fludarabine or alemtuzumab therapy. Patients who previously responded (complete response or partial response) to fludarabine or alemtuzumab therapy, but who have relapsed at the time of study entry, may be eligible but response to fludarabine or alemtuzumab therapy must have lasted >12 months (i.e., >12 months from a documented response to a documented relapse).
* Binet stage A, stage B, or stage C or Rai Stage I through IV disease with evidence of progression as evidenced by the presence of one or more of the following:

I. Evidence of progressive marrow failure as manifested by: 1) a decrease in hemoglobin to <11g/dL, or 2) a decrease in platelet count to <100 x 10^9/L within the previous 6 months, or 3) a decrease in absolute neutrophil count (ANC) to <1.0 X 10^9/L.

II. Progressive splenomegaly to >2 cm below the left costal margin or other organomegaly.

III. Progressive lymphadenopathy.

IV. Progressive lymphocytosis with an increase of 50% over a 2-month period, or an anticipated doubling time of less than 6 months.

* World Health Organization (WHO) performance status (PS) of 0 or 1.
* Life expectancy >12 weeks.
* Anti-cancer therapy, major surgery, or irradiation was completed >3 weeks before randomization in this study. Patient must have recovered from the acute side effects incurred as a result of previous therapy.
* Serum creatinine less than or equal to 2.0 x institutional upper limits of normal (ULN) and calculated creatinine clearance (CrCl) greater than or equal to 30mL/min using the Cockroft and Gault formula.
* Adequate liver function as indicated by a total bilirubin, AST, and ALT less than or equal to 2 x the institutional ULN value, unless directly attributable to the patient's tumor.
* Female patients with childbearing potential must have a negative serum pregnancy test with 2 weeks of first dose of study drug(s). Male and female patients must agree to use an effective contraceptive method while on study treatment, if appropriate, and for a minimum of 6 months following study therapy.
* Signed, written informed consent.

Exclusion Criteria:

* Previously treated with >1 prior regimen for B-CLL.
* Previously treated with a fludarabine plus alemtuzumab (FluCAM) regimen for B-CLL.
* Positive Coombs test and actively hemolyzing.
* Absolute neutrophil count (ANC) <1.5 x 10^9/L or platelet count <75 x 10^9/L, unless due to bone marrow involvement.
* Medical condition requiring chronic use of pharmacologic doses of oral corticosteroids, i.e. anything other than replacement dose levels.
* History of anaphylaxis following exposure to monoclonal antibodies.
* Use of investigational agents within 6 weeks prior to study randomization.
* Active infection or history of severe infection (grade 4) within 3 months prior to study randomization.
* Known to be human immunodeficiency virus (HIV) positive.
* Autoimmune thrombocytopenia.
* Active second malignancy.
* Known central nervous system (CNS) involvement with B-CLL.
* Other severe, concurrent diseases, including tuberculosis, mental disorders, serious cardiac functional capacity (Class III or IV as defined by the New York Heart Association Classification), severe diabetes, severe hypertension, pulmonary disease (chronic obstructive pulmonary disease [COPD] with hypoxemia), or major organ malfunction (liver, kidney) that could interfere with the patient's ability to participate in the study.
* Pregnant or nursing women.
* Patients that have progressed with more aggressive B-cell cancers such as Richter's syndrome.
* Active hepatitis or a history of prior viral hepatitis B or hepatitis C, or positive hepatitis B serologies without prior immunization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2004-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (48):
- Florida Cancer Specialists, Fort Myers, Florida, United States
- Austria (2):
  - Medizinische Universitatsklinik Graz, Graz
  - Universitat Wien AKH, Innere Medizin I, Vienna
- Bulgaria (5):
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski, Pleven
  - UMHAT St. Georgi, Hematology Clinic, Plovdiv
  - Multiprofile Hospital for Active Treatment "Alexandrovska", Sofia
  - National Center for Heamtology and Transfusiology, Sofia
  - Multiprofile Hospital for Active Treatment, St. Marina, Varna
- Canada (2):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
- Croatia (3):
  - Clinical Hospital Center Rijeka, Department of Haematology, Rijeka
  - Clinical Hospital Merkur, Zagreb
  - University Hospital Dubrava, Zagreb
- CHRU - Hopital Claude Huriez, Lille, France
- Germany (4):
  - Charite-Universitatsmedizin Berlin Campus Benjamin-Franklin, Berlin
  - Charite Universitatsklinikum der Humboldt-Universitat zu Berlin, Berlin
  - Klinikum der Universitat zu Koln, Klinik 1 fur Innere Medizin, Cologne
  - Robert-Bosch Krankenhaus GmbH, Stuttgart
- "Laikon" General Hospital, University of Athens, Goudi, Athens, Greece
- Italy (3):
  - U.O. Oncologia Medica Azienda Ospedaliera "Pugliese-Ciaccio", Cantanzaro
  - Unita Operativa di Medicina Generale Reumatologia e Oncoematologia, Milan
  - Istituto di Ematologia Dipartmento di Biotechnologie Celluari ed Ematologia, Universita di Roma "La Sapienza", Rome
- Poland (5):
  - Klinika Hematologii i Transplantacji Szpiku, Katowice
  - Klinika Hematologii AM, Lodz
  - Klinika Hematologii Pomorskiej Akademii Medycznej w Szczecinie, Szczecin
  - Katedra i Klinika Hamatologii, Onkologii I Chorob Wewnetrznych AM, Warsaw
  - Klinika Hematologii, Nowotworow Krwii 1 Transplantacji Szpiku, Wroclaw
- Portugal (2):
  - Hospital de Santa Maria Servico de Hematologia Clinica/Hospital de dia de Hematologia, Lisbon
  - Hospital de Sao Teotonio, Servico de Hematologia/Hosptial de Dia Oncologico, Viseu
- Institutol Clinic Fundeni, Clinica Heamtologie, Bucharest, Romania
- Russia (4):
  - GU "Main Military Clinical Hospital named after acad. N.N.Burdenko of MO of Russia", Haematology Centre 3, Moscow
  - GOUVPO "Saint-Petersburg State Medical University named after acad I.P.Pavlov of Roszdrav", Bone Marrow Transplantology Clinic, Saint Petersburg
  - Saint-Petersburg GUZ "City Hospital #31" 3, Dynamo Prospect, Saint Petersburg
  - State Healthcare Department "Sverdlovsk Regional Clinical Hospital #1",, Yekaterinburg
- Sweden (5):
  - University Hospital, Dept. of Hematology, Lund
  - Orebro University Hospital, Dep. of Medicine, Örebro
  - Universitetssjukhuset, Örebro
  - Medicin kliniken/Hematologsektionen, Sundsvall
  - Akademiska sjukhuset, Uppsala
- Ukraine (9):
  - Cherkasskly Oncology Dispensary, Cherkasy
  - City Clinical Hospital #4, Regional Hematology Center, Dnipro
  - Donetsk State Medical University, Donetsk
  - Kharkov Regional Clinical Oncology Center, Department of Hematology, Kharkiv
  - Khmelnitskiy Regional Hospital, Hematology Department, Khmelnitskiy
  - Institute of Oncology AMS of Ukraine, Kiev
  - Institute of Hematology and Transfusiology AMS of Ukraine, City Clinical Hospital #9, Kiev
  - Scientific Centre for Radiation Medicine AMS of Ukraine, Dept of Hematology and Transplantology, Kyiv
  - Lviv National Medical University named Danilo Galytcky, Lviv

REFERENCES:
- [Result] Engert A, et al. Overall Survival Advantage and Acceptable Safety Profile with Fludarabine in Combination with Alemtuzumab (FluCam) in Previously Treated Patients with Advanced Stage Chronic Lymphocytic Leukemia. Poster Presentation at American Society of Hematology 10 December 2010; Blood (ASH Annual Meeting Abstracts), Nov 2010;116:919. http://ash.confex.com/ash/2010/webprogram/Paper31687.html
- [Result] Engert A, et al. Improved Progression-free Survival (PFS) of Alemtuzumab (Campath®, MabCampath®) plus Fludarabine (Fludara®) versus Fludarabine Alone as Second-line Treatment of Patients with B-Cell Chronic Lymphocytic Leukemia: Preliminary Results from a Phase III Randomized Trial. 51st ASH Annual Meeting. Blood 2009;114. Abstract 537. http://ash.confex.com/ash/2009/webprogram/Paper21929.html
- [Result] Engert A, et al. Fludarabine (FLU) plus Alemtuzumab (FluCAM) Improves Progression Free Survival versus Fludarabine in Previously Treated Chronic Lymphocytic Leukemia and Demonstrates Activity in High Risk Patients. Poster Presentation at European Hematology Association 12 June 2010. Abstract 0768. http://www.eventure-online.com/eventure/publicAbstractView.do?id=136964&congressId=3446
- [Derived] Elter T, Gercheva-Kyuchukova L, Pylylpenko H, Robak T, Jaksic B, Rekhtman G, Kyrcz-Krzemien S, Vatutin M, Wu J, Sirard C, Hallek M, Engert A. Fludarabine plus alemtuzumab versus fludarabine alone in patients with previously treated chronic lymphocytic leukaemia: a randomised phase 3 trial. Lancet Oncol. 2011 Dec;12(13):1204-13. doi: 10.1016/S1470-2045(11)70242-X. Epub 2011 Oct 10. PMID 21992852

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment was from initiation of study drug(s) to 4 weeks after last administration of study drug. Follow-up was for those without disease progression and ended upon disease progression or primary endpoint analysis whichever came first. Observation included those with disease progression who were observed for alternative rx and overall survival.
Groups:
- Combination Arm (FluCAM): Participants received both fludarabine (Fludara) and alemtuzumab (Campath) intravenously. Initial escalation of alemtuzumab from 3 to 30 mg (escalation can take up to 14 days). Up to six cycles of fludarabine 30 mg/m^2 intravenous (IV) followed by alemtuzumab 30 mg IV on the first 3 days of each 28 day cycle.
- Fludarabine Alone: Participants received fludarabine monotherapy 25 mg/m^2 IV daily for the first 5 days of each 28 day cycle for up to 6 cycles.
Period: Treatment Period
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Started | 168 | 167
Safety Population | 164 (Four participants did not receive treatment) | 165 (Two participants did not receive treatment)
Completed | 103 (Finished 6 cycles of study drugs) | 107 (Finished 6 cycles of study drug)
Not Completed | 65 | 60
Not completed — Disease progression | 9 | 8
Not completed — Unable to comply with protocol | 3 | 1
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Physician Decision | 13 | 7
Not completed — AE - not treatment related | 7 | 7
Not completed — Toxicity - treatment related | 15 | 15
Not completed — Anemia or thrombocytopenia | 1 | 4
Not completed — Death | 5 | 7
Not completed — Other | 5 | 3
Period: Follow-up Period
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Started | 141 | 137
Completed | 37 | 18
Not Completed | 104 | 119
Not completed — Disease progression | 72 | 99
Not completed — Unable to comply with protocol | 5 | 0
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Physician Decision | 0 | 1
Not completed — AE - not related | 1 | 0
Not completed — Death | 13 | 7
Not completed — Other | 7 | 6
Period: Observation Period
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Started | 95 | 121
Completed | 49 | 56
Not Completed | 46 | 65
Not completed — Unable to comply with protocol | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Death | 33 | 55
Not completed — Other | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone | Total
Number analyzed (Participants) | 168 | 167 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (9.25) | 60.8 (9.34) | 60.4 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 59 | 118
  Male | 109 | 108 | 217
Race/Ethnicity, Customized [Number; unit: participants]
  White | 167 | 167 | 334
  Other | 1 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeters] | 169.0 (8.88) | 169.4 (9.30) | 169.2 (9.08)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: meters^2] | 1.87 (0.213) | 1.90 (0.218) | 1.88 (0.216)
Maximum Lymph Node Size [Number; unit: participants] — The number of participants whose largest lymph node by physical exam assessment during a baseline visit fell within two categories: <5 cm and >=5 cm. If there is no enlarged lymph node, then size is classified as <5 cm.
  participants
    <5 centimeters | 134 | 136 | 270
    >= 5 centimeters | 34 | 31 | 65
World Health Organization (WHO) Performance Status [Number; unit: participants] — Per protocol, all participants had a WHO performance status of 0 or 1. A WHO performance status of 0 is defined as "patient is able to carry out all normal activity without restriction," and status of 1 is "patient is ambulatory and capable of all self-care but unable to carry out any work; up and about more than 50% of waking hours."
  participants
    WHO Performance Status = 0 | 81 | 72 | 153
    WHO Performance Status = 1 | 87 | 95 | 182
Rai Stage Group [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity.
  Rai Stage 0: Lymphocytosis only, Rai Stage I: Lymphocytosis with lymphadenopathy, Rai Stage II: Lymphocytosis with hepatomegaly or splenomegaly, Rai Stage III: Lymphocytosis with anemia, Rai Stage IV: Lymphocytosis with thrombocytopenia.
  Per protocol, the 4 participants with Rai Stage 0 were eligible for the study because they had Binet Stage A.
  participants
    Rai Stage 0 | 2 | 2 | 4
    Rai Stage I - II | 104 | 102 | 206
    Rai Stage III - IV | 62 | 63 | 125
Binet Stage [Number; unit: participants] — Binet staging classifies CLL according to the number of lymphoid tissues involved, as well as the presence of low red blood cell count (anemia) or low number of blood platelets (thrombocytopenia).
  Binet Stage A: fewer than three areas of enlarged lymphoid tissue. Enlarged lymph nodes of the neck, underarms, and groin, as well as the spleen, are each considered "one group," whether unilateral (one-sided) or bilateral (on both sides).
  Binet Stage B: more than three areas of enlarged lymphoid tissue.
  Binet Stage C: anemia plus thrombocytopenia (platelets <100 x 10^3/dL).
  participants
    Binet Stage A | 27 | 25 | 52
    Binet Stage B | 89 | 89 | 178
    Binet Stage C | 52 | 53 | 105
Disease Status [Number; unit: participants] — Count of participants with refractory or relapsed disease at baseline (as reported by the investigator).
  participants
    Relapsed | 101 | 101 | 202
    Refractory | 67 | 66 | 133
Summary of Prior Therapy by Type of Therapy [Number; unit: participants] — Count of participants who had prior therapy categorized by type of therapy: fludarabine-containing therapy or non-fludarabine-containing therapy.
  participants
    Fludarabine-containing therapy | 25 | 26 | 51
    Non-fludarabine-containing therapy | 143 | 141 | 284

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Progression-free Survival (PFS) Based on Independent Response Review Panel (IRRP) Assessment
Description: Progression-free survival was defined as the number of days from the date of randomization to the date of first objective documentation of progressive disease (PD) as determined by the treatment-blinded IRRP, or death due to any cause. Results are expressed in months.
Time Frame: Up to 6 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
months | 23.65 [19.180 to 28.360] | 16.48 [12.500 to 21.220]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p < 0.001, Regression, Cox; Cox proportional hazards model was stratified by Rai Stage Group; Hazard Ratio (HR) = 0.610, 95% CI 2-sided [0.467 to 0.795]

2. Secondary Outcome: Participant Best Response to Treatment Assessed by the Independent Response Review Panel (IRRP)
Description: Participants were evaluated by the IRRP according to National Cancer Institute (NCI) 1996 response criteria. The best response observed during the study is summarized. Response categories include Complete Response (CR) with normal physical exam, marrow cells and blood values, Partial Response (PR) with a >= 50% decrease from baseline in lymphocytes, lymphadenopathy and liver or spleen exam, Stable Disease (SD) without significant progression from baseline, or Progressive Disease (PD) with increased size/number of nodes, size of liver or spleen, increase in lymphocytes, aggressive histology.
Time Frame: Up to 9 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
participants
  Overall Response (CR+PR) | 137 | 126
  Complete Response (CR) | 21 | 7
  Partial Response (PR) | 116 | 119
  Progressive Disease (PD) | 6 | 9
  Stable Disease (SD) | 12 | 21
  Not Evaluable (NE) | 13 | 11
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Comparison of Overall Response; Test type: Superiority or Other; p = 0.178, Cochran-Mantel-Haenszel — P-value presented is adjusted for multiple tests using Hochberg procedure for 3 clinically important secondary endpoints: ORR, CR rates and OS; CMH chi-square test for a difference in overall response rates between treatments stratified by Rai Stage Group; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.03 to 0.15] — Difference and confidence interval (CI) calculated using the recommended method by Altman et al
Statistical Analysis 2: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Comparison of complete response (CR); Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; CMH chi-square test for a difference in complete response rates between treatments stratified by Rai Stage Group; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.02 to 0.15] — Difference and confidence interval (CI) calculated using the recommended method by Altman et al

3. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival Time
Description: Overall survival was defined as the time in days from the date of randomization to the date of death due to any cause plus 1 day for all participants. Results are stated in months.
Time Frame: Up to 6 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
months | NA [NA to NA] — NA = values were not calculable since there were not enough events for the statistical estimation, ie, few participants died | 52.93 [40.890 to NA] — NA = values were not calculable since there were not enough events for the statistical estimation, ie, few participants died
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p = 0.042, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Cox proportional hazards model stratified by Rai Stage Group; Cox Proportional Hazard = 0.648, 95% CI 2-sided [0.449 to 0.937]

4. Secondary Outcome: Kaplan Meier Estimates for Time to Disease Progression Assessed by the Independent Response Review Panel (IRRP)
Description: Time to disease progression was defined as the number of days from the date of randomization to the date of first objective documentation of progressive disease as determined by IRRP. Results are stated in months.
Time Frame: Up to 6 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
months | 27.96 [22.340 to 31.910] | 18.68 [14.510 to 23.220]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p < 0.001, Regression, Cox; Cox regression model stratified by Rai Stage Group; Cox Proportional Hazard = 0.562, 95% CI 2-sided [0.420 to 0.752]

5. Secondary Outcome: Kaplan-Meier Estimates for Duration of Response Assessed by the Independent Response Review Panel (IRRP)
Description: Duration of response was analyzed for participants who achieved a complete response (CR) or partial response (PR) and was defined as the number of days from the first date of documented response to the date of progressive disease as determined by IRRP or death due to any cause. Results are stated in months.
Time Frame: Up to 6 years
Population: Full analysis set of participants who achieved a complete response or a partial response as determined by the IRRP.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 135 | 124
months | 25.10 [20.200 to 29.280] | 19.14 [14.140 to 21.910]

6. Secondary Outcome: Kaplan-Meier Estimates for Time to Alternative Therapy
Description: Time to alternative therapy was defined as the number of days from the date of randomization to the date of first alternative therapy for chronic lymphocytic leukemia (CLL) or death resulting from any cause. Participants who had not received alternative therapy as of the data cutoff date were censored at the last follow-up visit assessment date plus 1 day. Results are stated in months.
Time Frame: Up to 6 years
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
months | 25.43 [20.130 to 41.810] | 22.01 [20.130 to 27.830]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p = 0.021, Regression, Cox; Cox proportional hazards model stratified by Rai Stage Group; Cox Proportional Hazard = 0.718, 95% CI 2-sided [0.543 to 0.951]

7. Secondary Outcome: Mean EQ-5D™ Index Scores to Measure Quality of Life at Baseline
Description: EQ-5D™ is a trademark of the EuroQol Group. EQ-5D™ is a standardized instrument for use as a measure of health outcome. The questionnaire asks about health status along 5 dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression, which are rated at three possible levels (no problems, some problems, extreme problems). The score ranges from best (+1) to worst (-0.59).
Time Frame: Day 0 (baseline)
Population: Full analysis dataset. Participants who provided valid answers on questionnaires are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 164
units on a scale | 0.7959 (0.1868) | 0.7822 (0.2023)

8. Secondary Outcome: Mean EQ-5D™ Index Scores to Measure Quality of Life at End of Treatment
Description: as for outcome 7
Time Frame: up to month 6 (end of treatment)
Population: Full analysis dataset. Participants who provided valid answers on questionnaires are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 152 | 147
units on a scale | 0.8049 (0.2752) | 0.7749 (0.2569)

9. Secondary Outcome: Mean EuroQol Visual Analogue Scale (EQ-VAS) Scores to Measure Quality of Life at Baseline
Description: The EuroQol Visual Analogue Scale (EQ-VAS) was also used to capture the self-rating of current health status using a visual "thermometer" with the end points of 100 (best imaginable health state) at the top and zero (worst imaginable health state) at the bottom.
Time Frame: Day 0 (baseline)
Population: Full analysis set. Participants who provided valid answers on questionnaires are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 167 | 161
units on a scale | 70.9 (18.01) | 70.2 (17.24)

10. Secondary Outcome: Mean EuroQol Visual Analogue Scale (EQ-VAS) Scores to Measure Quality of Life at End of Treatment
Description: as for outcome 9
Time Frame: up to month 6 (end of treatment)
Population: Full analysis set. Participants who provided valid answers on questionnaires are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 152 | 146
units on a scale | 77.1 (19.41) | 75.7 (17.98)

11. Secondary Outcome: Summary of Participants With Adverse Experiences (AEs)
Description: Number of participants with adverse events (AEs). AEs were graded by the investigator using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and were assessed for relatedness to study treatment (4 point scale from 'not related' to 'definitely related'). Categories reported include participant counts for treatment-emergent AEs, AEs for infections, serious AEs, AEs causing discontinuation of study drug(s), and deaths. Related AEs for the combination arm can be related to either fludarabine or alemtuzumab.
Time Frame: Up to 6 years
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 164 | 165
participants
  At least 1 treatment emergent AE | 161 | 149
  At least 1 related treatment emergent AE | 159 | 125
  At least 1 treatment-emergent infection | 67 | 58
  At least 1 drug-related infection | 44 | 30
  At least 1 serious AE | 54 | 41
  At least 1 related serious AE | 47 | 28
  Discontinuation of study drug due to AE | 37 | 32
  Discontinuation of study drug due to related AE | 32 | 24
  Deaths | 10 | 12
  Patients who died due to a related AE | 7 | 6
  Patients who died within 30 days of the last dose | 4 | 7

12. Secondary Outcome: Mean Systemic Clearance (CL) of Fludarabine
Description: Clearance of drug from plasma is affected by the absorption, distribution, metabolism and elimination of the drug. Mean systemic clearance of fludarabine is derived from plasma concentration versus time data.
Time Frame: month 4 (cycle 4): first day of dosing (pre-dose, 0.5 hr end of infusion), second day of dosing (pre-dose, 0.5 hr end of infusion), third day of dosing (pre-dose, 0.25 hr, 0.5 hr end of infusion, 1,2,3,4,6,24,48,72 hr after start of fludarabine infusion)
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: liters/hour
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 17 | 12
liters/hour | 9.46 (4.31) | 9.54 (3.10)

13. Secondary Outcome: Total Volume of Distribution (Vss) of Fludarabine
Description: The total volume of distribution (Vss) is the apparent volume in which fludarabine is distributed immediately after it has been injected intravenously and equilibrated between plasma and the surrounding tissues. Total volume of distribution (Vss) of fludarabine is derived from plasma concentration versus time data.
Time Frame: as for outcome 12
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 17 | 12
liters | 117 (64.3) | 172 (91.3)

14. Other Pre Specified Outcome: Kaplan-Meier Estimates for Progression-free Survival (PFS) Based on Independent Response Review Panel (IRRP) for Participants With Rai Stage I-II
Description: Progression-free survival was defined as the number of days from the date of randomization to the date of first objective documentation of progressive disease (PD) as determined by the treatment-blinded IRRP, or death due to any cause. Results are expressed in months and include participants with Rai stage I or II.
Time Frame: Up to 6 years
Population: Full analysis set of participants with Rai stage I or II
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 104 | 102
months | 23.75 [19.970 to 29.700] | 20.76 [14.700 to 24.340]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p = 0.102, Regression, Cox; Cox Proportional Hazard = 0.750, 95% CI 2-sided [0.531 to 1.059]

15. Other Pre Specified Outcome: Kaplan-Meier Estimates for Progression-free Survival (PFS) Based on Independent Response Review Panel (IRRP) for Participants With Rai Stage III-IV
Description: Progression-free survival was defined as the number of days from the date of randomization to the date of first objective documentation of progressive disease (PD) as determined by the treatment-blinded IRRP, or death due to any cause. Results are expressed in months and include participants with Rai stage III or IV.
Time Frame: Up to 6 years
Population: Full analysis set of participants with Rai stage III or IV
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 62 | 63
months | 20.53 [14.310 to 31.910] | 11.51 [8.980 to 14.670]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p < 0.001, Regression, Cox; Cox Proportional Hazard = 0.443, 95% CI 2-sided [0.292 to 0.671]

16. Other Pre Specified Outcome: Kaplan-Meier Estimates of Overall Survival Time for Participants With Rai Stage I-II
Description: Overall survival was defined as the time in days from the date of randomization to the date of death due to any cause plus 1 day for all participants. Results are stated in months and include participants with Rai Stage I or II.
Time Frame: Up to 6 years
Population: Full analysis set of participants with Rai Stage I or II
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 104 | 102
months | NA [58.420 to NA] — NA=values were not calculable since there were not enough events for the statistical estimation, ie, few participants died | NA [57.430 to NA] — NA=values were not calculable since there were not enough events for the statistical estimation, ie, few participants died
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p = 0.819, Regression, Cox; Cox proportional hazards model; Cox Proportional Hazard = 1.066, 95% CI 2-sided [0.619 to 1.836]

17. Other Pre Specified Outcome: Kaplan-Meier Estimates of Overall Survival Time for Participants With Rai Stage III-IV
Description: Overall survival was defined as the time in days from the date of randomization to the date of death due to any cause plus 1 day for all participants. Results are stated in months and include participants with Rai Stage III or IV.
Time Frame: Up to 6 years
Population: Full analysis set of participants with Rai Stage III or IV
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 62 | 63
months | NA [32.140 to NA] — NA=values were not calculable since there were not enough events for the statistical estimation, ie, few participants died | 23.52 [17.760 to 40.300]
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p < 0.001, Regression, Cox; Cox proportional hazards model; Cox Proportional Hazard = 0.416, 95% CI 2-sided [0.250 to 0.690]

18. Secondary Outcome: Area Under the Curve (AUC) of Fludarabine From (AUC 0-tau)
Description: AUC (0-tau) is the area under the plasma concentration curve for fludarabine over the dosage interval (tau).
Time Frame: as for outcome 12
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 17 | 12
ng*h/mL | 8203 (6531) | 5669 (3888)

19. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Fludarabine
Description: Cmax is the maximum plasma concentration of fludarabine observed.
Time Frame: as for outcome 12
Population: Pharmacokinetic population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 17 | 12
ng/mL | 4084 (6089) | 1847 (1637)

20. Secondary Outcome: Participants With Minimal Residual Disease (MRD)
Description: MRD negativity in this report was defined by the absence of tumor cells in bone marrow, using 4-color flow cytometry. MRD was assessed in participants with a clinical complete response (CR) or partial response (PR) without recovery of blood counts. MRD represents a very positive outcome.
Time Frame: up to 9 months
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Number analyzed (Participants) | 168 | 167
participants | 6 | 0
Statistical Analysis 1: Comparison: Combination Arm (FluCAM) vs Fludarabine Alone; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel; CMH chi-square test for a difference in response rates between treatments stratified by Rai Stage Group; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [0.01 to 0.08]

ADVERSE EVENTS:
Time Frame: Up to 6 years
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Combination Arm (FluCAM) | Fludarabine Alone
Serious Adverse Events (participants affected / at risk) | 54/164 | 41/165
Other Adverse Events (participants affected / at risk) | 160/164 | 147/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Arm (FluCAM) (N=164) | Fludarabine Alone (N=165)
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 2 | 2
Autoimmune neutropenia (Blood and lymphatic system disorders) | 1 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 7
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 8 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Retinopathy (Eye disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 1
Sudden cardiac death (General disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1
Eye infection toxoplasmal (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Gastroenteritis escherichia coli (Infections and infestations) | 0 | 1
Hepatitis c (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci infection (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 2
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Cd4 lymphocytes decreased (Investigations) | 1 | 0
Cytomegalovirus test positive (Investigations) | 3 | 0
Pneumocystis test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Coma hepatic (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Radicular pain (Nervous system disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Arm (FluCAM) (N=164) | Fludarabine Alone (N=165)
Anaemia (Blood and lymphatic system disorders) | 36 | 39
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Granulocytopenia (Blood and lymphatic system disorders) | 3 | 1
Haematotoxicity (Blood and lymphatic system disorders) | 0 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 73 | 25
Lymphopenia (Blood and lymphatic system disorders) | 35 | 7
Neutropenia (Blood and lymphatic system disorders) | 82 | 84
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 44 | 44
Angina pectoris (Cardiac disorders) | 0 | 2
Aortic valve calcification (Cardiac disorders) | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 3
Pericardial effusion (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Accessory spleen (Congenital, familial and genetic disorders) | 1 | 0
Kidney malformation (Congenital, familial and genetic disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1
Goitre (Endocrine disorders) | 2 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 4
Diarrhoea (Gastrointestinal disorders) | 15 | 11
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 3
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingivitis ulcerative (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 3 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 20 | 13
Pancreatic disorder (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 4 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 15 | 3
Asthenia (General disorders) | 4 | 6
Catheter site inflammation (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 49 | 2
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 10 | 9
Generalised oedema (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 2 | 0
Hyperthermia (General disorders) | 6 | 0
Impaired healing (General disorders) | 0 | 1
Influenza like illness (General disorders) | 2 | 0
Infusion related reaction (General disorders) | 20 | 0
Injection site extravasation (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 0
Localised oedema (General disorders) | 0 | 3
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 6 | 4
Pyrexia (General disorders) | 96 | 14
Soft tissue inflammation (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 5 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis chronic active (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 7 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 5 | 1
Mycotic allergy (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Ascariasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 15 | 5
Bronchopneumonia (Infections and infestations) | 2 | 0
Bullous impetigo (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Folliculitis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 2 | 1
Herpes zoster (Infections and infestations) | 4 | 3
Infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 8
Neutropenic infection (Infections and infestations) | 2 | 1
Oral fungal infection (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 3 | 3
Otitis media (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 6 | 5
Pneumonia (Infections and infestations) | 6 | 3
Pulpitis dental (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 4 | 5
Respiratory tract infection viral (Infections and infestations) | 4 | 2
Rhinitis (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 1 | 3
Skin candida (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 3
Tooth infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 3 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 6 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 2
Beta 2 microglobulin decreased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatinine increased (Investigations) | 4 | 3
Blood lactate dehydrogenase increased (Investigations) | 3 | 0
Body temperature increased (Investigations) | 2 | 1
Breath sounds abnormal (Investigations) | 0 | 1
Cd4 lymphocytes decreased (Investigations) | 4 | 2
Creatinine renal clearance decreased (Investigations) | 5 | 5
Cytomegalovirus test positive (Investigations) | 19 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 2
Haemoglobin decreased (Investigations) | 4 | 5
Hepatic enzyme increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 6 | 7
Neutrophil pelger-huet anomaly present (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 6 | 10
Urine uric acid increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 2
Weight increased (Investigations) | 1 | 2
White blood cell count decreased (Investigations) | 7 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Fluid retention (Metabolism and nutrition disorders) | 2 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hyperproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic pemphigus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 5
Dysaesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Facial neuralgia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 14 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Radicular pain (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Sphenopalatine neuralgia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Crystalluria (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephroptosis (Renal and urinary disorders) | 2 | 0
Pollakiuria (Renal and urinary disorders) | 5 | 3
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Calculus prostatic (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 13 | 4
Drug eruption (Skin and subcutaneous tissue disorders) | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4
Pruritus allergic (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 25 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 22 | 4
Urticaria vesiculosa (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriosclerosis obliterans (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 11 | 6
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 2
Phlebitis (Vascular disorders) | 2 | 0
Systolic hypertension (Vascular disorders) | 1 | 1
Temporal arteritis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after an independent multi-investigator publication (in which the PI can participate) or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.